CLINICAL TRIAL: NCT01619475
Title: A2ALL: Adult-to-Adult Living Transplant Cohort Study
Brief Title: Adult-to-Adult Living Donor Transplant Cohort Study
Acronym: A2ALL-2
Status: Completed | Type: Observational
Sponsor: Arbor Research Collaborative for Health (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: A2ALL Core Protocol; U01DK085587 (NIH); U01DK085563 (NIH); U01DK085515 (NIH); U01DK062536 (NIH); U01DK062531 (NIH); U01DK062498 (NIH); U01DK062494 (NIH); U01DK062483 (NIH); U01DK062467 (NIH); U01DK062444 (NIH); 5U01DK062498-09 (NIH)
Record Dates: First submitted 2011-10-05; First posted 2012-06-14 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Liver Diseases; Hepatocellular Cancer; End Stage Liver Disease; Hepatitis C; Liver Cirrhosis
Keywords: Living Donor; Liver Transplantation; Quality of Life; Biosamples; Liver Recipient
MeSH Terms: conditions — Liver Diseases; Liver Neoplasms; End Stage Liver Disease; Hepatitis C; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — To collect biosamples prior to, during, and after LDLT among all donors and recipients. These biosamples include, liver biopsy,whole blood for genetic studies and DNA extraction, plasma, serum and peripheral cells to be retained in the bio-repository.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Prospective: Individuals approved as liver donors and recipients shortly Pre-donation/Pre-transplant at the study sites.
- Long-Term Follow-up: Donors and recipients enrolled in the original A2ALL Cohort study.
  Donors and LDLT recipients whose donation/transplant occurred during the period of time that began with the end of enrollment into the original Cohort study (Aug. 31, 2009) and ended with the opening of the enrollment in the current core protocol; this is referred to as the "Gap Era."
  LDLT recipients and donors who were not in the original Cohort study or from the Gap Era will enter the study at time proximate to time of living donation.
- HCV-Infected Liver Transplant Recipients: Male and female HCV-infected adult liver transplant recipients from those enrolled in the A2ALL-1 Cohort study and from those concurrently transplanted at the new A2ALL-2 centers (University of Toronto, University of Pittsburgh, Lahey Clinic).

SUMMARY:
The study is being conducted for the following reasons:

1. To determine the prevalence, course, and predictors of poor Health Related Quality of Life (HRQOL) outcomes associated with living donor donation.
2. To collect data and biosamples prior to, during, and after a living donor liver transplant (LDLT) among all donors and recipients for use by other adult-to-adult living donor liver transplant studies and future studies.
3. To study the effects of pressure and flow on the outcomes of LDLT.
4. To characterize the differences between living donor liver transplant and deceased donor liver transplant in terms of recipient post-transplant outcomes including patient and graft survival, surgical morbidity, and resource utilization.
5. To compare the long-term histological outcomes in recipients of LDLT and deceased donor liver transplant (DDLT) with recurrent hepatitis C virus (HCV) infection.
6. To understand the history of pain management and to measure quality of care in pain control in living donors following partial hepatectomy.

DETAILED DESCRIPTION:
The procedure of adult-to-adult living donor liver transplant (LDLT) is an extraordinary surgical therapy that involves the removal of 70% of the volume mass of an adult donor liver and its implantation into an adult recipient. A critical shortage of deceased donor livers, resulting in premature mortality among candidates in need of liver transplantation, remained the single most compelling force driving the need for adult-to-adult LDLT. Patients awaiting living donor liver transplant will be asked to enroll in this protocol at the time of identification of a potential living liver donor. Donors identified for the living donation will also be asked to enroll in the protocol. Donors and recipients who have already participated in a liver donation/transplant will be approached to join the protocol based on their clinical history.

Optimizing donors' health-related quality of life is a foremost goal for liver donor liver transplant programs and an overarching aim for this study. The proposed A2ALL-2 Health Related Quality of Life (HRQOL) Sub-Study will build upon the A2ALL HRQOL measures employed to date. There is a critical need to look at the important difficulties that liver donors appear to face not only in the early years but in the long-term after donation. Individuals who have enrolled in the study and are going to donate a portion of their liver will complete a HRQOL battery of tests conducted over the phone by experienced staff at Northwestern University or the University of Pittsburgh. The tests are a series of questions given to the upcoming donor at baseline (prior to the liver donation), at Month 3, and Month 6, Year 1 and Year 2 following donation. The new donor will complete up to 5 interviews by the survey research team. Individuals who have already donated (long-term donors), and out three years since donation can be enrolled, but they have to have donated in 2002 or more recently. Long-term follow-up donors will complete up to 4 interviews by the survey research team.

As LDLT moved from children to adults, it was observed early that the size of the graft was related to function in the recipient and that inadequate graft volume led to poor recipient outcomes. It has been found, that when the graft of the liver is too small, then the recipient can develop a number of symptoms including persistent ascites (fluid in the abdomen) and the graft becomes resistant to the passage of blood. This study hopes to develop and validate approaches that permit successful use of smaller donor livers and this is the principal goal of the surgical innovations portion of the study. The study will use standard surgical technique for the donor and recipient. Either right or left lobe donation and transplantation will be performed based on clinical parameters for graft selection.

Biosample collection of serum aliquots and liver tissue samples will be collected from subjects during different timepoints in the study. The collection of patient biosamples and DNA samples provides a resource with which researchers can rapidly validate clinical hypotheses and algorithms for clinical decision making. The collections also advance the development of diagnostic and prognostic markers and therapeutics. In addition, collection and storage of DNA samples may increase the sample size and the resulting power of a study to identify genetic determinants of a disease. The samples will be stored in the National Institute of Diabetic, Digestive and Kidney diseases (NIDDK) Repositories.

Hepatic C virus (HCV) recurrence after liver transplantation is universal in patients who have the virus pre-operatively. Chronic hepatitis evolves to a cirrhosis at a variable rate, but more rapidly than in non-transplant patients. The study will evaluate whether risk factors for aggressive HCV recurrence after DDLT also apply to LDLT recipients in long-term follow-up.

Pain control in living donors following partial hepatectomy will be measured as quality of care. The transplant community has no objective information about pain management in live liver donors to use for quality improvement. A validated tool to measure quality of pain management will be used to assess multidimensional aspects of pain care.

The following details the schedule of visits and the tests/procedures to be performed at each visit:

Recipient (before the surgery)

* Provide blood samples for the NIDDK Biosample Repository.
* Undergo imaging studies either Computed Assisted Tomography (CAT) or a Magnetic Resonance Imaging (MRI) to measure the size of the liver and spleen.
* If one has liver cancer or hepatocellular carcinoma (HCC), information will be collected about the tumor(s) and treatment.

Recipient (day of surgery)

* Provide a sample of the new liver to the NIDDK Biosample Repository.
* Provide blood samples immediately before and during the transplant surgery to the NIDDK Biosample Repository.
* Allow the researchers to collect information about the transplant surgery.
* Allow the researchers to collect information about any complications that develop after the transplant.
* During the transplant operation, an ultrasound probe will be applied to the two vessels going to the transplanted liver and a measurement of how much blood flows through these vessels to the liver will be taken. After less than 5 minutes the probe will be removed. Additionally, measurements will be taken of the pressure in one of the vessels, the portal vein, with a very small needle inserted by the surgeon. These measurements will be recorded and analyzed as part of the study.
* During living donor transplant surgery, it is occasionally necessary to adjust the blood flow to the liver to improve the function. If the surgeon determines that the flow to the liver needs to be adjusted, the measurements described above will be repeated after the adjustments have been made. These measurements will be recorded and analyzed as part of the study.
* Additional tests which are standard of care may also be carried out at the site.
* If one has HCC,then information will be collected about the tumor(s).

Recipient(immediately after the surgery)

* Provide blood samples during the first and second weeks after the transplant to the NIDDK Biosample Repository.
* Allow the researchers to collect information about the lab tests (liver function tests, blood counts,etc.).
* Undergo an ultrasound measurement of the blood flow through the portal vein on the day after the operation.
* Additional tests which are standard of care may be also carried out at the site.

Recipient (throughout the course of the study)

* Provide blood samples to the NIDDK Biosample Repository at months 1, 3, and 12, and annually thereafter though August 2014. Approximately 10 teaspoons or 50 ccs of blood will be collected at each assessment.
* Undergo imaging studies at three months after the operation (either a CAT or MRI) of the liver and spleen to see how much the liver has grown since the transplant operation.
* Return to the transplant center for assessment at months 1,3, and 12, and annually thereafter through August 2014.
* Allow the researchers to collect information about any hospitalizations that occur after the transplant operation.
* Allow the researchers to collect information about any complications that develop after the transplant, through August 2014.
* Allow the researchers to collect information about any liver biopsies that are performed after the transplant.
* If the subject has Hepatitis C (HCV) and is post-transplant, and has had a liver transplant from a living donor or a deceased donor, the subject will be asked permission for review of the chart and collect information about the pre-transplant HCV treatment, the transplant operation, the immunosuppression medications, rejection episodes, and any HCV treatment received prior to consenting to this study.
* If the subject has HCV,and has given permission, the chart will be reviewed for liver biopsy results that occurred at least three years after the transplant.
* If a liver biopsy was not done at least three years after the transplant or if the recent liver biopsy was at least three years after the transplant but the most recent liver biopsy was more than one year the subject will be a asked to come to the center and get a liver biopsy done.
* If the study liver biopsy is done, or information on a previous biopsy has been collected the slides of the liver tissue obtained will be sent to the central pathologist to read. The name of the subject and any other identifying information will not be on the slides. It will have a code number on it that links back to the subject's clinical data.
* If the HCV subject is unwilling or unable to undergo a liver biopsy, then the subject will be asked to undergo a procedure called "transient elastography". Transient elastography is a non-invasive procedure during which a sound wave is transmitted to the liver through an ultrasound probe, and the time it takes for the sound wave to travel through the liver is measured. Transient elastography is considered to be an experimental procedure. However, it has been well-studied, and there have been no adverse events or injuries with its use.
* If the subject has HCV, some blood will be collected for storage in the NIDDK Repository. Approximately 10 teaspoons or 50ccs of blood will be collected at that time.

Donor (before the surgery)

* The subject will be called on the telephone by the survey researchers to answer questions about health, and well-being as well as views about the donation process.
* The survey questions may take up to 45 minutes to complete.
* Provide blood cell samples for the NIDDK Biosample Repository. Approximately 12 teaspoons or 60 ccs of blood will be collected.
* Undergo an imaging study before the operation (either CAT or MRI) to measure the size of the liver and spleen.
* Additional tests which are standard of care may also be carried out at the site.

Donor (day of the surgery)

* Provide samples of liver to the NIDDK Biosample Repository.
* Allow the researchers to collect information about the donation surgery.
* Allow the researchers to collect information about any complications that develop after the donation.

Donor (immediately after the surgery)

* Two days after the surgery, the subject will be asked questions about their post-operative pain.
* Provide blood samples one week after the donation surgery to the NIDDK Biosample Repository. Approximately 5-6 teaspoons or 25-30ccs of blood will be collected.

Donor (throughout the course of the study)

* Provide blood samples to the NIDDK Biosample Repository at week 1, month 1, month 3, and month 12. Approximately 10 teaspoons or 50 ccs of blood will be collected at each assessment.
* Return to the transplant center for assessment at month 3, and annually thereafter through August 2014.
* Undergo an imaging study at three months after the operation (CAT or MRI) to measure the size of the liver and spleen to see how much the liver has grown back since the donation operation.
* If the subject entered this study prior to undergoing surgery, questions will have to be answered by telephone about quality of life after donation at 3, 6, 12, and 24 months following donation. These telephone interviews may take up to 45 minutes to complete.
* If the subject entered the study after living liver donation, questions will be asked over the telephone about quality of life upon study entry and then annually for three years. The telephone interviews may take 45 minutes to complete.
* Allow the researchers to collect information about any complications that develop after the donation operation, through August 2014.
* Allow the researchers to collect information about the hospitalizations that occur after the transplant operation.

ELIGIBILITY:
Inclusion Criteria:

Recipients

1. Age 18 or older at the time of consent
2. Has had a living donor identified and accepted and LDLT is planned
3. Informed consent obtained
4. Is listed for single organ (liver) transplantation

Donors

1. Age 18 or older at the time of consent
2. Has undergone donor evaluation process and was accepted and donation surgery is planned
3. Informed consent obtained

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The sample population will consist of the following:
  * Donors and LDLT and DDLT recipients enrolled in the original A2ALL cohort study.
  * Donors and LDLT recipients where the donation/transplant occurred during the period of time that began with the end of enrollment into the original Cohort study (August 31, 2009) and ended with the opening of enrollment in the current core protocol; this is referred to as the "Gap Era."
  * Prospective donors and LDLT recipients for donation/transplant surgery.
  * HCV-infected adult liver transplant recipients enrolled in the A2ALL-1 Cohort and from those currently transplanted at the new A2ALL-2 centers (University of Toronto, University of Pittsburgh, and Lahey Clinic).
Sampling Method: Non-Probability Sample
Enrollment: 1871 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Recipient patient and graft survival starting from the time of transplantation in LDLT & DDLT. | Yearly follow-up starting at transplant, measured between enrollment and up to 4 years.
  To characterize the differences between LDLT and DDLT in terms of recipient post-transplant outcomes for patient and graft survival.
Number and severity of surgical complications and resource utilization after transplant. | Yearly follow-up starting at transplant, measured between enrollment , and up to 4 years.
  Comparison of incidence of defined medical and surgical complications after transplant between LDLT and DDLT.
  Comparison of resource utilization (hospitalization) between LDLT and DDLT.
Health Related Quality of Life (HRQOL) in living liver donors. | Yearly assessment from donation up to 5 assessments.
  To estimate the prevalence, course, and predictors of poor HRQOL outcomes associated with living liver donation.
Number of Blood/Tissue Samples from Donors and Recipients. | Yearly samples starting at transplant/donation (donors until year 1, and recipients until year 4.)
  To collect data and biosamples prior to, during, and after LDLT among all donors and recipients for use by other A2ALL protocols and future studies.
Pressure and Flow Measurements during the transplant surgery in LDLT recipients. | During the transplant (at completion of dissection, and after revascularization).
  To establish normal hepatic blood flow and portal compliance in the human liver, to examine the relationships among hepatic flow and pressure, graft size and function, and clinical outcomes.
Measures of liver fibrosis (Ishak score) in LDLT and DDLT recipients with recurrent HCV infection. | Enrollment up to 4 years, with data collected at the time of each liver biopsy.
  To assess whether recurrent Hepatitis C is histologically less severe in LDLT compared with DDLT recipients.
Pain control in living donors following partial hepatectomy | The first 48 hours after donation surgery
  Self-reported pain and satisfaction with pain management during the first 48 hours after donation surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Merion, MD, Study Chair — University of Michigan; Averell Sherker, MD, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (9):
- United States (8):
  - University of California, San Francisco, California
  - University of Colorado Health Sciences, Aurora, Colorado
  - Northwestern University, Division of Transplantation, Chicago, Illinois
  - Lahey Clinic, Burlington, Massachusetts
  - Columbia University, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Virginia Commonwealth University-Medical College of Virginia, Richmond, Virginia
- University of Toronto, Toronto, Ontario, Canada

REFERENCES:
- [Background] Olthoff KM, Merion RM, Ghobrial RM, Abecassis MM, Fair JH, Fisher RA, Freise CE, Kam I, Pruett TL, Everhart JE, Hulbert-Shearon TE, Gillespie BW, Emond JC; A2ALL Study Group. Outcomes of 385 adult-to-adult living donor liver transplant recipients: a report from the A2ALL Consortium. Ann Surg. 2005 Sep;242(3):314-23, discussion 323-5. doi: 10.1097/01.sla.0000179646.37145.ef. PMID 16135918
- [Background] Freise CE, Gillespie BW, Koffron AJ, Lok AS, Pruett TL, Emond JC, Fair JH, Fisher RA, Olthoff KM, Trotter JF, Ghobrial RM, Everhart JE; A2ALL Study Group. Recipient morbidity after living and deceased donor liver transplantation: findings from the A2ALL Retrospective Cohort Study. Am J Transplant. 2008 Dec;8(12):2569-79. doi: 10.1111/j.1600-6143.2008.02440.x. Epub 2008 Oct 24. PMID 18976306
- [Background] Trotter JF, Hill-Callahan MM, Gillespie BW, Nielsen CA, Saab S, Shrestha R, Talamantes MM, Weinrieb RM; A2ALL Study Group. Severe psychiatric problems in right hepatic lobe donors for living donor liver transplantation. Transplantation. 2007 Jun 15;83(11):1506-8. doi: 10.1097/01.tp.0000263343.21714.3b. PMID 17565325
- [Background] Trotter JF, Wisniewski KA, Terrault NA, Everhart JE, Kinkhabwala M, Weinrieb RM, Fair JH, Fisher RA, Koffron AJ, Saab S, Merion RM; A2ALL Study Group. Outcomes of donor evaluation in adult-to-adult living donor liver transplantation. Hepatology. 2007 Nov;46(5):1476-84. doi: 10.1002/hep.21845. PMID 17668879
- [Background] Terrault NA, Shiffman ML, Lok AS, Saab S, Tong L, Brown RS Jr, Everson GT, Reddy KR, Fair JH, Kulik LM, Pruett TL, Seeff LB; A2ALL Study Group. Outcomes in hepatitis C virus-infected recipients of living donor vs. deceased donor liver transplantation. Liver Transpl. 2007 Jan;13(1):122-9. doi: 10.1002/lt.20995. PMID 17192908
- [Background] Fisher RA, Kulik LM, Freise CE, Lok AS, Shearon TH, Brown RS Jr, Ghobrial RM, Fair JH, Olthoff KM, Kam I, Berg CL; A2ALL Study Group. Hepatocellular carcinoma recurrence and death following living and deceased donor liver transplantation. Am J Transplant. 2007 Jun;7(6):1601-8. doi: 10.1111/j.1600-6143.2007.01802.x. PMID 17511683
- [Background] Campsen J, Blei AT, Emond JC, Everhart JE, Freise CE, Lok AS, Saab S, Wisniewski KA, Trotter JF; Adult-to-Adult Living Donor Liver Transplantation Cohort Study Group. Outcomes of living donor liver transplantation for acute liver failure: the adult-to-adult living donor liver transplantation cohort study. Liver Transpl. 2008 Sep;14(9):1273-80. doi: 10.1002/lt.21500. PMID 18756453
- [Background] Ghobrial RM, Freise CE, Trotter JF, Tong L, Ojo AO, Fair JH, Fisher RA, Emond JC, Koffron AJ, Pruett TL, Olthoff KM; A2ALL Study Group. Donor morbidity after living donation for liver transplantation. Gastroenterology. 2008 Aug;135(2):468-76. doi: 10.1053/j.gastro.2008.04.018. Epub 2008 Apr 22. PMID 18505689
- [Background] Shaked A, Ghobrial RM, Merion RM, Shearon TH, Emond JC, Fair JH, Fisher RA, Kulik LM, Pruett TL, Terrault NA; A2ALL Study Group. Incidence and severity of acute cellular rejection in recipients undergoing adult living donor or deceased donor liver transplantation. Am J Transplant. 2009 Feb;9(2):301-8. doi: 10.1111/j.1600-6143.2008.02487.x. Epub 2008 Dec 15. PMID 19120082
- [Background] Trotter JF, Gillespie BW, Terrault NA, Abecassis MM, Merion RM, Brown RS Jr, Olthoff KM, Hayashi PH, Berg CL, Fisher RA, Everhart JE; Adult-to-Adult Living Donor Liver Transplantation Cohort Study Group. Laboratory test results after living liver donation in the adult-to-adult living donor liver transplantation cohort study. Liver Transpl. 2011 Apr;17(4):409-17. doi: 10.1002/lt.22246. PMID 21445924
- [Background] Olthoff KM, Abecassis MM, Emond JC, Kam I, Merion RM, Gillespie BW, Tong L; Adult-to-Adult Living Donor Liver Transplantation Cohort Study Group. Outcomes of adult living donor liver transplantation: comparison of the Adult-to-adult Living Donor Liver Transplantation Cohort Study and the national experience. Liver Transpl. 2011 Jul;17(7):789-97. doi: 10.1002/lt.22288. PMID 21360649
- [Result] Berg CL, Gillespie BW, Merion RM, Brown RS Jr, Abecassis MM, Trotter JF, Fisher RA, Freise CE, Ghobrial RM, Shaked A, Fair JH, Everhart JE; A2ALL Study Group. Improvement in survival associated with adult-to-adult living donor liver transplantation. Gastroenterology. 2007 Dec;133(6):1806-13. doi: 10.1053/j.gastro.2007.09.004. Epub 2007 Sep 14. PMID 18054553
- [Result] Abecassis MM, Fisher RA, Olthoff KM, Freise CE, Rodrigo DR, Samstein B, Kam I, Merion RM; A2ALL Study Group. Complications of living donor hepatic lobectomy--a comprehensive report. Am J Transplant. 2012 May;12(5):1208-17. doi: 10.1111/j.1600-6143.2011.03972.x. Epub 2012 Feb 15. PMID 22335782
- [Result] Berg CL, Merion RM, Shearon TH, Olthoff KM, Brown RS Jr, Baker TB, Everson GT, Hong JC, Terrault N, Hayashi PH, Fisher RA, Everhart JE. Liver transplant recipient survival benefit with living donation in the model for endstage liver disease allocation era. Hepatology. 2011 Oct;54(4):1313-21. doi: 10.1002/hep.24494. PMID 21688284
- [Result] Butt Z, Dew MA, Liu Q, Simpson MA, Smith AR, Zee J, Gillespie BW, Abbey SE, Ladner DP, Weinrieb R, Fisher RA, Hafliger S, Terrault N, Burton J, Sherker AH, DiMartini A. Psychological Outcomes of Living Liver Donors From a Multicenter Prospective Study: Results From the Adult-to-Adult Living Donor Liver Transplantation Cohort Study2 (A2ALL-2). Am J Transplant. 2017 May;17(5):1267-1277. doi: 10.1111/ajt.14134. Epub 2017 Jan 3. PMID 27865040
- [Result] Dew MA, DiMartini AF, Ladner DP, Simpson MA, Pomfret EA, Gillespie BW, Merion RM, Zee J, Smith AR, Holtzman S, Sherker AH, Weinrieb R, Fisher RA, Emond JC, Freise CE, Burton JR Jr, Butt Z. Psychosocial Outcomes 3 to 10 Years After Donation in the Adult to Adult Living Donor Liver Transplantation Cohort Study. Transplantation. 2016 Jun;100(6):1257-69. doi: 10.1097/TP.0000000000001144. PMID 27152918
- [Result] DiMartini AF, Dew MA, Butt Z, Simpson MA, Ladner DP, Smith AR, Hill-Callahan P, Gillespie BW. Patterns and predictors of sexual function after liver donation: The Adult-to-Adult Living Donor Liver Transplantation Cohort study. Liver Transpl. 2015 May;21(5):670-82. doi: 10.1002/lt.24108. PMID 25779554
- [Result] DiMartini A, Dew MA, Liu Q, Simpson MA, Ladner DP, Smith AR, Zee J, Abbey S, Gillespie BW, Weinrieb R, Mandell MS, Fisher RA, Emond JC, Freise CE, Sherker AH, Butt Z. Social and Financial Outcomes of Living Liver Donation: A Prospective Investigation Within the Adult-to-Adult Living Donor Liver Transplantation Cohort Study 2 (A2ALL-2). Am J Transplant. 2017 Apr;17(4):1081-1096. doi: 10.1111/ajt.14055. Epub 2016 Nov 10. PMID 27647626
- [Result] Emond JC, Fisher RA, Everson G, Samstein B, Pomposelli JJ, Zhao B, Forney S, Olthoff KM, Baker TB, Gillespie BW, Merion RM. Changes in liver and spleen volumes after living liver donation: a report from the Adult-to-Adult Living Donor Liver Transplantation Cohort Study (A2ALL). Liver Transpl. 2015 Feb;21(2):151-61. doi: 10.1002/lt.24062. PMID 25488878
- [Result] Emond JC, Goodrich NP, Pomposelli JJ, Baker TB, Humar A, Grant DR, Abt P, Friese CE, Fisher RA, Kam I, Sherker AH, Gillespie BW, Merion RM. Hepatic Hemodynamics and Portal Flow Modulation: The A2ALL Experience. Transplantation. 2017 Oct;101(10):2375-2384. doi: 10.1097/TP.0000000000001823. PMID 28514251
- [Result] Everson GT, Hoefs JC, Niemann CU, Olthoff KM, Dupuis R, Lauriski S, Herman A, Milne N, Gillespie BW, Goodrich NP, Everhart JE. Functional elements associated with hepatic regeneration in living donors after right hepatic lobectomy. Liver Transpl. 2013 Mar;19(3):292-304. doi: 10.1002/lt.23592. PMID 23239552
- [Result] Everson GT, Terrault NA, Lok AS, Rodrigo del R, Brown RS Jr, Saab S, Shiffman ML, Al-Osaimi AM, Kulik LM, Gillespie BW, Everhart JE; Adult-to-Adult Living Donor Liver Transplantation Cohort Study. A randomized controlled trial of pretransplant antiviral therapy to prevent recurrence of hepatitis C after liver transplantation. Hepatology. 2013 May;57(5):1752-62. doi: 10.1002/hep.25976. Epub 2013 Jan 17. PMID 22821361
- [Result] Gillespie BW, Merion RM, Ortiz-Rios E, Tong L, Shaked A, Brown RS, Ojo AO, Hayashi PH, Berg CL, Abecassis MM, Ashworth AS, Friese CE, Hong JC, Trotter JF, Everhart JE; A2ALL Study Group. Database comparison of the adult-to-adult living donor liver transplantation cohort study (A2ALL) and the SRTR U.S. Transplant Registry. Am J Transplant. 2010 Jul;10(7):1621-33. doi: 10.1111/j.1600-6143.2010.03039.x. Epub 2010 Feb 25. PMID 20199501
- [Result] Gordon FD, Goldberg DS, Goodrich NP, Lok AS, Verna EC, Selzner N, Stravitz RT, Merion RM. Recurrent primary sclerosing cholangitis in the Adult-to-Adult Living Donor Liver Transplantation Cohort Study: Comparison of risk factors between living and deceased donor recipients. Liver Transpl. 2016 Sep;22(9):1214-22. doi: 10.1002/lt.24496. Epub 2016 Aug 2. PMID 27339253
- [Result] Kulik LM, Fisher RA, Rodrigo DR, Brown RS Jr, Freise CE, Shaked A, Everhart JE, Everson GT, Hong JC, Hayashi PH, Berg CL, Lok AS; A2ALL Study Group. Outcomes of living and deceased donor liver transplant recipients with hepatocellular carcinoma: results of the A2ALL cohort. Am J Transplant. 2012 Nov;12(11):2997-3007. doi: 10.1111/j.1600-6143.2012.04272.x. Epub 2012 Sep 20. PMID 22994906
- [Result] Ladner DP, Dew MA, Forney S, Gillespie BW, Brown RS Jr, Merion RM, Freise CE, Hayashi PH, Hong JC, Ashworth A, Berg CL, Burton JR Jr, Shaked A, Butt Z. Long-term quality of life after liver donation in the adult to adult living donor liver transplantation cohort study (A2ALL). J Hepatol. 2015 Feb;62(2):346-53. doi: 10.1016/j.jhep.2014.08.043. Epub 2014 Sep 6. PMID 25195558
- [Result] Levitsky J, Goldberg D, Smith AR, Mansfield SA, Gillespie BW, Merion RM, Lok AS, Levy G, Kulik L, Abecassis M, Shaked A. Acute Rejection Increases Risk of Graft Failure and Death in Recent Liver Transplant Recipients. Clin Gastroenterol Hepatol. 2017 Apr;15(4):584-593.e2. doi: 10.1016/j.cgh.2016.07.035. Epub 2016 Aug 25. PMID 27567694
- [Result] Mandell MS, Smith AR, Dew MA, Gordon DB, Holtzman S, Howell T, DiMartini AF, Butt Z, Simpson MA, Ladner DP, Freise CE, McCluskey SA, Fisher RA, Guarrera JV, Olthoff KM, Pomfret EA. Early Postoperative Pain and its Predictors in the Adult to Adult Living Donor Liver Transplantation Cohort Study. Transplantation. 2016 Nov;100(11):2362-2371. doi: 10.1097/TP.0000000000001442. PMID 27517726
- [Result] Merion RM, Shearon TH, Berg CL, Everhart JE, Abecassis MM, Shaked A, Fisher RA, Trotter JF, Brown RS Jr, Terrault NA, Hayashi PH, Hong JC; A2ALL Study Group. Hospitalization rates before and after adult-to-adult living donor or deceased donor liver transplantation. Ann Surg. 2010 Mar;251(3):542-9. doi: 10.1097/SLA.0b013e3181ccb370. PMID 20130466
- [Result] Olthoff KM, Emond JC, Shearon TH, Everson G, Baker TB, Fisher RA, Freise CE, Gillespie BW, Everhart JE. Liver regeneration after living donor transplantation: adult-to-adult living donor liver transplantation cohort study. Liver Transpl. 2015 Jan;21(1):79-88. doi: 10.1002/lt.23966. Epub 2014 Oct 6. PMID 25065488
- [Result] Olthoff KM, Smith AR, Abecassis M, Baker T, Emond JC, Berg CL, Beil CA, Burton JR Jr, Fisher RA, Freise CE, Gillespie BW, Grant DR, Humar A, Kam I, Merion RM, Pomfret EA, Samstein B, Shaked A. Defining long-term outcomes with living donor liver transplantation in North America. Ann Surg. 2015 Sep;262(3):465-75; discussion 473-5. doi: 10.1097/SLA.0000000000001383. PMID 26258315
- [Result] Pomposelli JJ, Goodrich NP, Emond JC, Humar A, Baker TB, Grant DR, Fisher RA, Roberts JP, Olthoff KM, Gillespie BW, Merion RM. Patterns of Early Allograft Dysfunction in Adult Live Donor Liver Transplantation: The A2ALL Experience. Transplantation. 2016 Jul;100(7):1490-9. doi: 10.1097/TP.0000000000001240. PMID 27326811
- [Result] Samstein B, Smith AR, Freise CE, Zimmerman MA, Baker T, Olthoff KM, Fisher RA, Merion RM. Complications and Their Resolution in Recipients of Deceased and Living Donor Liver Transplants: Findings From the A2ALL Cohort Study. Am J Transplant. 2016 Feb;16(2):594-602. doi: 10.1111/ajt.13479. Epub 2015 Oct 13. PMID 26461803
- [Result] Terrault NA, Stravitz RT, Lok AS, Everson GT, Brown RS Jr, Kulik LM, Olthoff KM, Saab S, Adeyi O, Argo CK, Everhart JE, Rodrigo del R; A2ALL Study Group. Hepatitis C disease severity in living versus deceased donor liver transplant recipients: an extended observation study. Hepatology. 2014 Apr;59(4):1311-9. doi: 10.1002/hep.26920. Epub 2014 Mar 1. PMID 24677192
- [Result] Zimmerman MA, Baker T, Goodrich NP, Freise C, Hong JC, Kumer S, Abt P, Cotterell AH, Samstein B, Everhart JE, Merion RM. Development, management, and resolution of biliary complications after living and deceased donor liver transplantation: a report from the adult-to-adult living donor liver transplantation cohort study consortium. Liver Transpl. 2013 Mar;19(3):259-67. doi: 10.1002/lt.23595. PMID 23495079